CLINICAL TRIAL: NCT07148557
Title: A Single-center, Open-label, Phase Ib Clinical Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Characteristics of LP-003 Injection in Adolescent Subjects Aged 12-18 Years
Brief Title: A Study of Single Dose of LP-003 in Adolescent Subjects
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P10-LP003-09
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Spontaneous Urticaria (CSU); Seasonal Allergic Rhinitis (SAR)
MeSH Terms: conditions — Chronic Urticaria; Rhinitis, Allergic, Seasonal | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: LP-003 Dose 1 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 1 (Single)
- Cohort 2 : LP-003 Dose 2 (Single) (Experimental)
  Interventions: Biological: LP-003 Dose 2 (Single)

INTERVENTIONS:
Biological: LP-003 Dose 1 (Single) — A single dose of LP-003 (400 mg/dose) was SC
  Arms: Cohort 1: LP-003 Dose 1 (Single)
Biological: LP-003 Dose 2 (Single) — A single dose of LP-003 (600 mg/dose) was SC
  Arms: Cohort 2 : LP-003 Dose 2 (Single)

SUMMARY:
This is a single-center, open-label, phase Ib clinical study to evaluate the safety, pharmacokinetics and pharmacodynamic characteristics of LP-003 injection in adolescent subjects aged 12-18 years.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent subjects aged ≥12 years and <18 years, male or female.
* History of allergic diseases (self-reported is acceptable), including, but not limited to, food allergies, allergic rhinitis, allergic asthma, urticaria, and atopic dermatitis.
* Agreement to use effective contraception during the study and for 6 months after the end of the study.
* Subject and parent or legal guardian able to understand and voluntarily sign the informed consent form, and comply with study visits and related procedures.

Exclusion Criteria:

* Allergic to LP-003 or its excipients.
* Any serious or uncontrolled chronic disease (e.g., severe arrhythmia, ischemic heart disease, NYHA Class III/IV heart failure, severe pulmonary disease, inadequately controlled asthma, hypertension, diabetes, hypo- or hyperthyroidism) that may affect subject safety as determined by the Investigator.
* History of severe allergic reactions.
* Abnormal venous access, venipuncture or subcutaneous injection intolerance, history of needle or blood phobia.
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m² at screening.
* ALT or AST > ULN and considered clinically significant by the Investigator.
* Any other abnormal screening test result that, in the Investigator's opinion, could affect subject safety or study assessments.
* Systemic corticosteroid therapy (intravenous, intramuscular, or oral) within 4 weeks prior to study drug administration.
* Use of medications known to interact with epinephrine (e.g., β-blockers, ACE inhibitors, tricyclic antidepressants) within 4 weeks prior to administration.
* Use of biologic products (e.g., omalizumab) within 6 months prior to administration.
* Receipt vaccines within 14 days before administration or planning vaccination during the study.
* Participation in other clinical trials within 3 months prior to screening or within 5 half-lives of investigational product discontinuation (whichever is longer).
* Any other conditions that the Investigator considers subjects unsuitable for participation in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Observation for 196 days after administration
  Number of subjects with treatment-related Treatment Emergent Adverse Events (TEAEs).

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) of LP-003 | Observation for 196 days after administration
  The time when the blood drug concentration reaches its peak after a single dose of medication.
Maximum concentration (Cmax) of LP-003 | Observation for 196 days after administration
  The maximum concentration of LP-003 in the bloodstream after administration.
Elimination half-life (t1/2) of LP-003 | Observation for 196 days after administration
  The time required for the concentration of LP-003 in the bloodstream to decrease by half.
Area under the concentration-time curve (AUC0-t) of LP-003 | Observation for 196 days after administration
  The area under the concentration-time curve (AUC) from time zero to the last chosen time point represents the integral of the drug concentration in the bloodstream over the specified duration.
Apparent clearance rate (CL/F) of LP-003 | Observation for 196 days after administration
  The ratio of drug clearance to drug concentration, represents the apparent clearance of a drug after administration, adjusted for bioavailability.
Assessment of total immunoglobulin E (IgE) | Observation for 196 days after administration
  The changes in serum total IgE levels compared to baseline at different assessment time points.
Assessment of free immunoglobulin E (IgE) | Observation for 196 days after administration
  The changes in serum free IgE levels compared to baseline at different assessment time points.
Assessment of immunogenicity | Observation for 196 days after administration
  The proportion of anti drug antibody (ADA) positive subjects at different detection time points.

IPD SHARING:
Plan to Share IPD: No